CLINICAL TRIAL: NCT07039669
Title: A Multi-Centered, Randomized, Double-Blinded, Placebo-Controlled Phase III Clinical Trial, to Evaluate the Efficacy and Safety of 611 in Chinese Adults With Moderate to Severe Chronic Obstructive Pulmonary Disease
Brief Title: Evaluation of 611 in Chinese Adults Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSGJ-611-COPD-III-01
Record Dates: First submitted 2025-06-05; First posted 2025-06-26 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive (COPD)
MeSH Terms: conditions — Lung Diseases; Pulmonary Disease, Chronic Obstructive | interventions — entacapone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 611 (Experimental): 611 Q2W, subcutaneous (SC) injection
  Interventions: Drug: 611
- placebo (Placebo Comparator): placebo Q2W, subcutaneous (SC) injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 611 — 611 subcutaneous (SC) injection
  Arms: 611
Drug: Placebo — placebo Q2W, subcutaneous (SC) injection
  Arms: placebo

SUMMARY:
The objective of the study was to evaluate the efficacy and safety of 611 in Chinese adults with moderate to severe COPD.

DETAILED DESCRIPTION:
The maximum study duration was 66 weeks per participants, including a screening period of up to 6 weeks, a 52-week randomized treatment period, and a 8-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and follow the protocol requirements, and give written informed consent prior to participation voluntarily in the study.
2. Male or female adults ages 40 to 85 years old when signing the informed consent.
3. Current or former smokers with a smoking history of ≥10 pack-years.
4. Documented diagnosis of COPD for at least 12 months prior to enrolment
5. Moderate-to-severe COPD.
6. Documented history of ≥ 2 moderate or ≥ 1 severe COPD exacerbations within 12 months prior to enrolment.
7. Background triple therapy (ICS + LABA + LAMA) for 3 months prior to randomization with a stable dose of medication for ≥ 1 month prior to randomization; Double therapy (LABA + LAMA) allowed if ICS is contraindicated.
8. Female subjects of reproductive age (and their male partners) and male subjects (and their female partners) must use highly effective contraception throughout the study period and for at least 3 months after the last dose. The subjects had no plans to pregnancy, donate sperm or donate egg during the whole study period and for at least 3 months after the last dose.

Exclusion Criteria:

1. Presence of a known pre-existing, clinically important lung condition other than COPD.
2. A current diagnosis of asthma or history of asthma according to the Global Initiative for Asthma (GINA) guidelines or other accepted guidelines.
3. Diagnosis of α-1 anti-trypsin deficiency.
4. Presence of an active autoimmune disease.
5. Subjects who have any malignant tumors within 5 years prior to enrollment.
6. Known, pre-existing other concurrent clinically significant medical conditions that are uncontrolled.
7. Diagnosed active parasitic infection, suspected or high risk of parasitic infection.
8. Subjects who have active Hepatitis B, Hepatitis C or HIV infections as determined by positive results at Screening.
9. Known with allergic or intolerant to any biological product.
10. Any reason which, in the opinion of investigator, would prevent the subject from participating in the study.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 594 (Estimated)
Dates: Start 2025-07-16 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Annualized rate of moderate or severe COPD Exacerbations | Baseline to Week 52
  Moderate exacerbations were recorded by the Investigator and defined as acute exacerbation of COPD (AECOPD) event that required systemic corticosteroids with/without antibiotics. Severe exacerbations were also recorded by the Investigator and defined as AECOPD event that required hospitalization or observation for >24 hours in an emergency department/urgent care facility or resulted in death.

SECONDARY OUTCOMES:
Change from baseline in pre-bronchodilator FEV1 at Week 24 | Baseline, Week 24
  FEV1 is the Forced expiratory volume in one second at study site
Time to first Moderate or severe COPD exacerbation | Baseline to Week 52
  Moderate exacerbations were recorded by the Investigator and defined as acute exacerbation of COPD (AECOPD) event that required systemic corticosteroids with/without antibiotics. Severe exacerbations were also recorded by the Investigator and defined as AECOPD event that required hospitalization or observation for >24 hours in an emergency department/urgent care facility or resulted in death.
Annualized rate of severe COPD Exacerbations | Baseline to Week 52
  Severe exacerbations were recorded by the Investigator and defined as AECOPD event that required hospitalization or observation for >24 hours in an emergency department/urgent care facility or resulted in death.
Change from baseline in pre-bronchodilator FEV1 | Baseline to Week 52
  FEV1 is the Forced expiratory volume in one second at study site
Change from baseline in SGRQ scores | Baseline to Week 52
  St. George's Respiratory Questionnaire (SGRQ).The SGRQ is a 50-item self-administered questionnaire designed to measure and quantify health status in adult participants with chronic airflow limitation. Scores by dimension were calculated for 3 domains: symptoms (respiratory symptoms: frequency and severity), activity (activities that cause or are limited by breathlessness) and impacts (social functioning and psychological disturbances due to airway disease). Total score was obtained by summing all positive responses in the questionnaire. The minimum and maximum values were 0 and 100, respectively. Higher scores mean a worse outcome. Baseline was defined as the last available value up to randomization but prior to the first dose of study treatment.
Percentage of participants with a decrease in SGRQ total score of ≥ 4 points from baseline | Baseline to Week 16
  Percentage of participants with a decrease in SGRQ total score of ≥ 4 points from baseline
Change from baseline in post-bronchodilator FEV1 | Baseline to Week 52
  FEV1 is the Forced expiratory volume in one second at study site
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs) | Up to 60 Weeks
  An AE was defined as any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An SAE was defined as any untoward medical occurrence that: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. TEAEs were defined as AEs that developed or worsened or became serious during TE period (between the first administration of study treatment to the last administration of the study treatment + 14 days).
611 Concentration in Serum | Baseline to Week 60
  The concentration of 611 in Serum
Percentage of Participants With Anti-drug Antibodies and Neutralizing Antibodies | Baseline to Week 60
  Immunogenicity assessment will be based on Anti-drug Antibodies (ADAs) response and development of Neutralizing Antibodies (NABs). Percentage is calculated based on the number of evaluable participants and was calculated by number of participants with treatment-emergent positive anti-drug antibodies / number of evaluable participants * 100%
Change in serum concentrations of Pulmonary and activation-regulated chemokine (PARC) | Baseline to Week 60
  Change in serum concentrations of PARC
Change in serum concentrations of IgE | Baseline to Week 60
  Change in serum concentrations of IgE

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - ZheJiang Provincial People's Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No